CLINICAL TRIAL: NCT04333797
Title: Multicentre Prospective Cohort Study Assessing Risk and Protective Factors to Develop Psychopathology in Transitional Age Youth
Brief Title: Psychiatry of Transition in a World in Transition
Acronym: Transition_psy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Erasme University Hospital (Other); Brugmann University Hospital (Other); Service santé mentale à l'ULB (Unknown); Université Libre de Bruxelles (Other); King Baudouin Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P2020/PSY/Transition_psy
Record Dates: First submitted 2020-03-27; First posted 2020-04-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2020-06

CONDITIONS: Transitional Care; Mental Disorder in Adolescence; Mental Health
Keywords: Transitional age youth; CAMHS; AMHS; Dimensional approach; Child and Adolescent Psychiatry services; Adult Psychiatry services
MeSH Terms: conditions — Psychological Well-Being | interventions — Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transitional age youth (Other): Assessed group.
  Interventions: Other: Risk and Protective Factors Assessment

INTERVENTIONS:
Other: Risk and Protective Factors Assessment — First assessment at baseline (T0) - 17 y.o. Follow-up 2 years later (T1) - 19 y.o.
  Other Names: Transitional care from CAMHS to AMHS

SUMMARY:
This clinical study evaluates risk and protective factor to develop psychopathology in transitional age youth. 300 patients will be recruited at the age of 17 years old and assessed at baseline and 2 years later.

DETAILED DESCRIPTION:
Emerging adults are a particularly at-risk population in mental health. Transitional age youth have specific needs, not currently covered between child and adolescent mental health services (CAMHS) and adult mental health services (AMHS), mainly because of existing barriers. Movements from one to the other must be planned to achieve optimal patient care.

Our project aims to identify clinical dimensional characteristics contributing to the development of psychopathology during the transition period. Continuities, discontinuities and resilience factors will be explored. The final purpose is to develop a non-stigmatizing approach to reduce rejection from youths in psychopathological suffering and increase social inclusion.

The transversal and trans-diagnostic approach consists of a dimensional evaluation: 300 youth at the age of 17 will be included in a cohort of in-patients, out-patients and control group. Participants will be assessed at baseline and 2 years later. The primary outcome is based on Health of the Nation Outcome Scale for Children and Adolescents, measuring mental health care need, and WHO Quality of Life assessment.

The secondary outcomes include the assessment of dimensions representing risk or protective factors to develop psychopathology and evolution of mental health status during transition age. Baseline evaluation consists in internalizing/externalizing symptoms, impulsivity/compulsivity, emotion regulation, cognitive functioning, social and family functioning, developmental, medical and trauma history. At follow-up, mental health pathways and transition results will be described.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking and French-understanding
* Subjects who accepted to participated to the study (signature of informed consent/assent document from subjects and parents or legal holder of parental authority)
* Specific criteria for patients: inpatients and out-patients
* Specific criteria for control group: youth from general population or placed in residential centres

Exclusion Criteria:

* Impossibility to answer to the assessment tools
* Medium intellectual disability (homogenous IQ < 75)
* Presence of a grave somatic disease (cancer, cardiac failure, renal failure, central nervous system disorder), that is progressive or that affects the vital prognosis in the short term
* Active participation to another study

Ages: 17 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline self-rated mental health status (need for care) at 2 years | Change from Baseline HoNOSCA before transition at 17 y.o. to after transition at 19 y.o.
  Measured at baseline (T0) and follow-up (T1) with the Health of the Nation Outcome Scale for Children and Adolescents (HoNOSCA).
Change from Baseline self-rated measure of quality of life at 2 years | Change from Baseline WHO-QoL before transition at 17 y.o. to after transition at 19 y.o
  Measured at baseline (T0) and follow-up (T1) with the Quality of life assessed by World Health Organisation Quality of Life Assessment (WHO-QoL-BREF)

SECONDARY OUTCOMES:
Self-rated measure of traumatic life events | Before transition at 17 y.o. (T0)
  Measured with Childhood Trauma Questionnaire (CTQ)
Self-rated measure of family functioning | Before transition at 17 y.o. (T0)
  Measured with Family Assessment Device (FAD)
Self-rated measure to quantify the risk of developing psychiatric disorders | Before transition at 17 y.o. (T0)
  Measured with General Health Questionnaire (GHQ-12)
Self-rated measure of internalising and externalising symptoms | Before transition at 17 y.o. (T0)
  Measured with Youth Self Report 11-18 (YSR)
Self-rated measure of impulsivity and compulsivity | Before transition at 17 y.o. (T0)
  Measured with Barratt Impulsiveness Scale (BIS-11)
Self-rated measure of depressivity | Before transition at 17 y.o. (T0)
  Measured with Beck Depression Inventory-II (BDI-II)
Self-rated measure of suicidal risk | Before transition at 17 y.o. (T0)
  Measured with Beck Scale of Suicide Ideation (BSS)
Self-rated measure of emotional regulation | Before transition at 17 y.o. (T0)
  Measured with Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA)
Self-rated measure of interpersonal relationships social adaptation | Before transition at 17 y.o. (T0)
  Measured with Social Adaptation Self-evaluation Scale (SASS)
Self-rated measure of cognitive insight | Before transition at 17 y.o. (T0)
  Measured with Beck Cognitive Insight Scale (BCIS)
Cognitive assessment - IQ | Before transition at 17 y.o. (T0)
  Measured with Wechsler Adult Intelligence Scale (WAIS-IV)
Executive functions assessment - alertness, divided attention, flexibility and working memory | Before transition at 17 y.o. (T0)
  Measured with Test of Attentional Performance (TAP)
Executive functions assessment - cognitive inhibition | Before transition at 17 y.o. (T0)
  Measured with STROOP Task
Executive functions assessment - planning task | Before transition at 17 y.o. (T0)
  Measured with Tower of London Test (TOL)
Self-rated measure of executive functions | Before transition at 17 y.o. (T0)
  Measured with Behavior Rating Inventory of Executive Function - Self report (BRIEF-SR)
Self-rated measure of transition readiness and appropriateness | Before transition at 17 y.o. (T0)
  Measured with Transition Readiness and Appropriateness Mesure (TRAM)
Self-rated measure of therapeutic alliance | After transition at 19 y.o. (T1)
  Measured with Helping Alliance Questionnaire (HAQ)
Self-rated measure of transition related outcomes | After transition at 19 y.o. (T1)
  Measured with Transition Related Outcomes Mesure (TROM)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Delvenne, MD, PhD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (4):
- Belgium (4):
  - Brugmann University Hospital, Brussels
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - Service santé mentale à l'ULB, Brussels
  - Erasme University Hospital, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caspi A, Moffitt TE. All for One and One for All: Mental Disorders in One Dimension. Am J Psychiatry. 2018 Sep 1;175(9):831-844. doi: 10.1176/appi.ajp.2018.17121383. Epub 2018 Apr 6. PMID 29621902
- [Background] Tuomainen H, Schulze U, Warwick J, Paul M, Dieleman GC, Franic T, Madan J, Maras A, McNicholas F, Purper-Ouakil D, Santosh P, Signorini G, Street C, Tremmery S, Verhulst FC, Wolke D, Singh SP; MILESTONE consortium. Managing the link and strengthening transition from child to adult mental health Care in Europe (MILESTONE): background, rationale and methodology. BMC Psychiatry. 2018 Jun 4;18(1):167. doi: 10.1186/s12888-018-1758-z. PMID 29866202
- [Background] Singh SP, Paul M, Ford T, Kramer T, Weaver T. Transitions of care from Child and Adolescent Mental Health Services to Adult Mental Health Services (TRACK Study): a study of protocols in Greater London. BMC Health Serv Res. 2008 Jun 23;8:135. doi: 10.1186/1472-6963-8-135. PMID 18573214
- [Background] Hovish K, Weaver T, Islam Z, Paul M, Singh SP. Transition experiences of mental health service users, parents, and professionals in the United Kingdom: a qualitative study. Psychiatr Rehabil J. 2012 Winter;35(3):251-7. doi: 10.2975/35.3.2012.251.257. PMID 22246124
- [Background] Leebens PK, Williamson ED. Developmental Psychopathology: Risk and Resilience in the Transition to Young Adulthood. Child Adolesc Psychiatr Clin N Am. 2017 Apr;26(2):143-156. doi: 10.1016/j.chc.2016.12.001. PMID 28314447
- [Background] Singh SP, Tuomainen H. Transition from child to adult mental health services: needs, barriers, experiences and new models of care. World Psychiatry. 2015 Oct;14(3):358-61. doi: 10.1002/wps.20266. No abstract available. PMID 26407794
- [Background] Paul M, Street C, Wheeler N, Singh SP. Transition to adult services for young people with mental health needs: A systematic review. Clin Child Psychol Psychiatry. 2015 Jul;20(3):436-57. doi: 10.1177/1359104514526603. Epub 2014 Apr 7. PMID 24711585
- [Background] McGorry P, Bates T, Birchwood M. Designing youth mental health services for the 21st century: examples from Australia, Ireland and the UK. Br J Psychiatry Suppl. 2013 Jan;54:s30-5. doi: 10.1192/bjp.bp.112.119214. PMID 23288499
- [Background] Gore FM, Bloem PJ, Patton GC, Ferguson J, Joseph V, Coffey C, Sawyer SM, Mathers CD. Global burden of disease in young people aged 10-24 years: a systematic analysis. Lancet. 2011 Jun 18;377(9783):2093-102. doi: 10.1016/S0140-6736(11)60512-6. Epub 2011 Jun 7. PMID 21652063
- [Background] Kotov R, Ruggero CJ, Krueger RF, Watson D, Yuan Q, Zimmerman M. New dimensions in the quantitative classification of mental illness. Arch Gen Psychiatry. 2011 Oct;68(10):1003-11. doi: 10.1001/archgenpsychiatry.2011.107. PMID 21969458
- [Background] Kim-Cohen J, Caspi A, Moffitt TE, Harrington H, Milne BJ, Poulton R. Prior juvenile diagnoses in adults with mental disorder: developmental follow-back of a prospective-longitudinal cohort. Arch Gen Psychiatry. 2003 Jul;60(7):709-17. doi: 10.1001/archpsyc.60.7.709. PMID 12860775
- [Background] Jones PB. Adult mental health disorders and their age at onset. Br J Psychiatry Suppl. 2013 Jan;54:s5-10. doi: 10.1192/bjp.bp.112.119164. PMID 23288502
- [Background] Snyder HR, Gulley LD, Bijttebier P, Hartman CA, Oldehinkel AJ, Mezulis A, Young JF, Hankin BL. Adolescent emotionality and effortful control: Core latent constructs and links to psychopathology and functioning. J Pers Soc Psychol. 2015 Dec;109(6):1132-49. doi: 10.1037/pspp0000047. Epub 2015 May 25. PMID 26011660
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Copeland WE, Wolke D, Shanahan L, Costello EJ. Adult Functional Outcomes of Common Childhood Psychiatric Problems: A Prospective, Longitudinal Study. JAMA Psychiatry. 2015 Sep;72(9):892-9. doi: 10.1001/jamapsychiatry.2015.0730. PMID 26176785
- [Background] Ormel J, Oerlemans AM, Raven D, Laceulle OM, Hartman CA, Veenstra R, Verhulst FC, Vollebergh W, Rosmalen JG, Reijneveld SA, Oldehinkel AJ. Functional outcomes of child and adolescent mental disorders. Current disorder most important but psychiatric history matters as well. Psychol Med. 2017 May;47(7):1271-1282. doi: 10.1017/S0033291716003445. Epub 2017 Jan 9. PMID 28065168
- [Background] Kessler RC, Amminger GP, Aguilar-Gaxiola S, Alonso J, Lee S, Ustun TB. Age of onset of mental disorders: a review of recent literature. Curr Opin Psychiatry. 2007 Jul;20(4):359-64. doi: 10.1097/YCO.0b013e32816ebc8c. PMID 17551351
- [Background] Paus T, Keshavan M, Giedd JN. Why do many psychiatric disorders emerge during adolescence? Nat Rev Neurosci. 2008 Dec;9(12):947-57. doi: 10.1038/nrn2513. Epub 2008 Nov 12. PMID 19002191
- [Background] Chatburn A, Coussens S, Kohler MJ. Resiliency as a mediator of the impact of sleep on child and adolescent behavior. Nat Sci Sleep. 2013 Dec 23;6:1-9. doi: 10.2147/NSS.S54913. eCollection 2013. PMID 24379734
- [Background] Andersen SL. Commentary on the special issue on the adolescent brain: Adolescence, trajectories, and the importance of prevention. Neurosci Biobehav Rev. 2016 Nov;70:329-333. doi: 10.1016/j.neubiorev.2016.07.012. Epub 2016 Jul 14. PMID 27423540
- [Background] Georgieff N. L'adolescence à l'épreuve de la neurobiologie ? Adolescence [Internet]. 2013;T.31 1(1):185. Available from: http://www.cairn.info/revue-adolescence-2013-1-page-185.htm
- [Background] National Institute of Mental Health. The Teen Brain: Still Under Construction. Natl Inst Ment Heal [Internet]. 2011;1-10. Available from: http://www.nimh.nih.gov/health/publications/the-teen-brain-still-under-construction/index.shtml
- [Background] Copeland W, Shanahan L, Costello EJ, Angold A. Cumulative prevalence of psychiatric disorders by young adulthood: a prospective cohort analysis from the Great Smoky Mountains Study. J Am Acad Child Adolesc Psychiatry. 2011 Mar;50(3):252-61. doi: 10.1016/j.jaac.2010.12.014. Epub 2011 Jan 26. PMID 21334565
- [Background] Lamb, C., Hall, D., Kelvin, R., & Van Beinum M. Working at the CAMHS/Adult Interface: Good practice guidance for the provision of psychiatric services to adolescents/young adults. London R Coll Psychiatr. 2008;
- [Background] Jivanjee, P., & Kruzich J. Supports for young people with mental health conditions and their families in the transition years. Best Pract Ment Health. 2011;7(1):115-33.
- [Background] Pottick KJ, Bilder S, Vander Stoep A, Warner LA, Alvarez MF. US patterns of mental health service utilization for transition-age youth and young adults. J Behav Health Serv Res. 2008 Oct;35(4):373-89. doi: 10.1007/s11414-007-9080-4. Epub 2007 Nov 17. PMID 18026842
- [Background] Blum RW, Garell D, Hodgman CH, Jorissen TW, Okinow NA, Orr DP, Slap GB. Transition from child-centered to adult health-care systems for adolescents with chronic conditions. A position paper of the Society for Adolescent Medicine. J Adolesc Health. 1993 Nov;14(7):570-6. doi: 10.1016/1054-139x(93)90143-d. No abstract available. PMID 8312295
- [Background] Singh SP, Paul M, Ford T, Kramer T, Weaver T, McLaren S, Hovish K, Islam Z, Belling R, White S. Process, outcome and experience of transition from child to adult mental healthcare: multiperspective study. Br J Psychiatry. 2010 Oct;197(4):305-12. doi: 10.1192/bjp.bp.109.075135. PMID 20884954
- [Background] Cosgrave EM, Yung AR, Killackey EJ, Buckby JA, Godfrey KA, Stanford CA, et al. Met and unmet need in youth mental health. J Ment Heal [Internet]. 2008 Jan 6;17(6):618-28. Available from: http://www.tandfonline.com/doi/full/10.1080/09638230701506267
- [Background] Singh SP. Transition of care from child to adult mental health services: the great divide. Curr Opin Psychiatry. 2009 Jul;22(4):386-90. doi: 10.1097/YCO.0b013e32832c9221. PMID 19417667
- [Background] Achenbach T. Youth Self-Report Form and Profile for Ages 11-18 (YSR/11-18). Itaca, Ill Riverside. 1991;
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Beck A, Steer R, Brown G. Beck depression inventory-II. San Antonio. 1996;78(2):490.
- [Background] Beck A, Steer R. BSS: Beck scale for suicide ideation. Psychol Corp. 1991;
- [Background] Gosling CJ, Noblecourt K, Moutier S. Questionnaire de régulation émotionnelle pour enfants et adolescents. Enfance. 2018;N°2(2):291.
- [Background] Goldberg D, Williams P. General health questionnaire (GHQ). Swindon, Wiltshire, UK nferNelson. 2000
- [Background] Gowers SG, Harrington RC, Whitton A, Lelliott P, Beevor A, Wing J, Jezzard R. Brief scale for measuring the outcomes of emotional and behavioural disorders in children. Health of the Nation Outcome Scales for children and Adolescents (HoNOSCA). Br J Psychiatry. 1999 May;174:413-6. doi: 10.1192/bjp.174.5.413. PMID 10616607
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Bernstein DP, Ahluvalia T, Pogge D, Handelsman L. Validity of the Childhood Trauma Questionnaire in an adolescent psychiatric population. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):340-8. doi: 10.1097/00004583-199703000-00012. PMID 9055514
- [Background] Epstein NB, Baldwin LM, Bishop DS. The McMaster Family Assessment Device. J Marital Fam Ther [Internet]. 1983 Apr;9(2):171-80. Available from: http://doi.wiley.com/10.1111/j.1752-0606.1983.tb01497.x
- [Background] Bosc M, Dubini A, Polin V. Development and validation of a social functioning scale, the Social Adaptation Self-evaluation Scale. Eur Neuropsychopharmacol. 1997 Apr;7 Suppl 1:S57-70; discussion S71-3. doi: 10.1016/s0924-977x(97)00420-3. PMID 9169311
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Singh SP, Tuomainen H, Girolamo G, Maras A, Santosh P, McNicholas F, Schulze U, Purper-Ouakil D, Tremmery S, Franic T, Madan J, Paul M, Verhulst FC, Dieleman GC, Warwick J, Wolke D, Street C, Daffern C, Tah P, Griffin J, Canaway A, Signorini G, Gerritsen S, Adams L, O'Hara L, Aslan S, Russet F, Davidovic N, Tuffrey A, Wilson A, Gatherer C, Walker L; MILESTONE Consortium. Protocol for a cohort study of adolescent mental health service users with a nested cluster randomised controlled trial to assess the clinical and cost-effectiveness of managed transition in improving transitions from child to adult mental health services (the MILESTONE study). BMJ Open. 2017 Oct 16;7(10):e016055. doi: 10.1136/bmjopen-2017-016055. PMID 29042376
- [Background] Wechsler D. Wechsler adult intelligence scale, 4th ed. San Antonio, TX Pearson. 2008
- [Background] Ryan JJ, Kreiner DS, Gontkovsky ST, Glass Umfleet L. Classification Accuracy of Sequentially Administered WAIS-IV Short Forms. Appl Neuropsychol Adult. 2015;22(6):409-14. doi: 10.1080/23279095.2014.953677. Epub 2015 Mar 18. PMID 25785485
- [Background] Zimmermann P, Fimm B. Tests d'évaluation de l'attention (TEA). Würselen: Psytest. 1994
- [Background] Stroop JR. Studies of interference in serial verbal reactions. J Exp Psychol [Internet]. 1935;18(6):643-62. Available from: http://content.apa.org/journals/xge/18/6/643
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Roussel M, Goldefroy O. La batterie GREFEX: données normatives. Fonct exécutives Pathol Neurol Psychiatr. 2008;231-52.
- [Background] Shallice T. Specific impairments of planning. Philos Trans R Soc Lond B Biol Sci. 1982 Jun 25;298(1089):199-209. doi: 10.1098/rstb.1982.0082. PMID 6125971
- [Background] Coyette F, Van der Linden M. Adaptation de l'Épreuve de la Tour de Londres. Unpubl Doc Cent Revalidation Neuropsychol des Clin Univ Saint-Luc, Bruxelles Serv Neuropsychol l'Université Liege, Belgium. 1993
- [Background] Gioia GA, Isquith PK. Behavior Rating Inventory for Executive Functions. In: Kreutzer JS, DeLuca J, Caplan B, editors. Encyclopedia of Clinical Neuropsychology [Internet]. New York, NY: Springer New York; 2011. p. 372-6. Available from: http://link.springer.com/10.1007/978-0-387-79948-3
- [Background] Kermarrec S, Kabuth B, Bursztejn C, Guillemin F. French adaptation and validation of the helping alliance questionnaires for child, parents, and therapist. Can J Psychiatry. 2006 Dec;51(14):913-22. doi: 10.1177/070674370605101407. PMID 17249634
- [Background] Luborsky L, Barber JP, Siqueland L, Johnson S, Najavits LM, Frank A, Daley D. The Revised Helping Alliance Questionnaire (HAq-II) : Psychometric Properties. J Psychother Pract Res. 1996 Summer;5(3):260-71. PMID 22700294
- [Derived] Marchini S, Reis J, Ben-Shaool E, Delhaye M, Kornreich C, Nicolis H, Slama H, Leys C, Delvenne V. Dimensional model on how familial vulnerability and environmental factors impact transitional age youth psychopathology: The Transition_psy study. Front Psychiatry. 2023 Mar 23;14:1103030. doi: 10.3389/fpsyt.2023.1103030. eCollection 2023. PMID 37032919
- [Derived] Reis J, Marchini S, De Leeuw A, Slama H, Leys C, Delhaye M, Kornreich C, Nicolis H, Delvenne V. Study Protocol: Transition_psy a Multicenter Prospective Longitudinal Cohort Study Assessing Risk and Protective Factors to Develop Psychopathology in Transitional Age Youth in Belgium. Front Psychiatry. 2021 Jun 21;12:645679. doi: 10.3389/fpsyt.2021.645679. eCollection 2021. PMID 34234697